CLINICAL TRIAL: NCT00445146
Title: A Phase 2, Open-Label, Multicenter Study of the Safety of Ritonavir-Boosted GS-9137 (GS-9137/r) Administered in Combination With Other Antiretroviral Agents for the Treatment of HIV-1 Infected Subjects
Brief Title: Safety of EVG+RTV Administered With Other Antiretroviral Agents for the Treatment of HIV-1 Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-183-0130
Record Dates: First submitted 2007-02-28; First posted 2007-03-08 (Estimated); Results first posted 2016-04-25 (Estimated); Last update posted 2016-04-25 (Estimated); Status verified 2016-03

CONDITIONS: HIV Infections
Keywords: Phase 2; Open-label; Rollover; Integrase Inhibitor; Antiretroviral Agents; Highly Active Antiretroviral Activity; HAART; HIV, HIV-1, AIDS virus, Human Immunodeficiency Virus; Acquired Immune Deficiency Syndrome Virus; treatment experienced
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — elvitegravir; Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- EVG+RTV (Experimental): EVG 85 mg or 150 mg + RTV + ARV regimen
  Participants receiving lopinavir/ritonavir (LPV/r) or atazanavir/ritonavir (ATV/r) as part of their ARV regimen will receive EVG 85 mg and all other participants will receive EVG 150 mg.
  Some participants may receive EVG 300 mg during the course of protocol amendment 2.
  Interventions: Drug: EVG; Drug: RTV; Drug: ARV regimen

INTERVENTIONS:
Drug: EVG — Elvitegravir (EVG) tablet administered orally once daily with food
  Other Names: Vitekta®; GS-9137
Drug: RTV — Ritonavir (RTV; /r) 100 mg capsule administered orally once daily with food
  Other Names: Norvir®
Drug: ARV regimen — The components of the ARV regimen will be selected by the investigator without input from the sponsor. The antiretroviral regimen must consist of at least 2 agents, not including the non-nucleoside reverse transcriptase inhibitors (NNRTIs) efavirenz, nevirapine, or delavirdine; the protease inhibitors saquinavir, nelfinavir, or indinavir; or investigational agents (without sponsor approval).

SUMMARY:
The main objective of this study is to observe the long-term safety of elvitegravir (EVG) boosted with ritonavir (RTV) in combination with other antiretroviral (ARV) agents in participants who have completed a prior EVG+RTV treatment study.

ELIGIBILITY:
Inclusion Criteria:

* Completion of a prior EVG+RTV treatment study without treatment-limiting toxicity.
* Males and females of childbearing potential must agree to utilize effective contraception methods.
* Ability to understand and sign a written informed consent form.

Exclusion Criteria:

* Females who are pregnant or breastfeeding.
* Participation in any other clinical trial without prior approval from the Sponsor.
* Any other clinical condition or prior therapy that, in the opinion of the investigator, would make the subject unsuitable for the study.
* Subjects receiving ongoing therapy with contraindicated drugs.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2007-02; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Rhee, MD, Study Director — Gilead Sciences
Locations (48):
- United States (47):
  - Pheonix, Arizona
  - Little Rock, Arkansas
  - Beverly Hills, California
  - Costa Mesa, California
  - Fountain Valley, California
  - Long Beach, California
  - Los Angeles, California
  - Newport Beach, California
  - Palo Alto, California
  - San Diego, California
  - San Francisco, California
  - Norwalk, Connecticut
  - Washington D.C., District of Columbia
  - Atlantis, Florida
  - Fort Lauderdale, Florida
  - Manors, Florida
  - Miami, Florida
  - North Miami Beach, Florida
  - North Palm Beach, Florida
  - Orlando, Florida
  - Sarasota, Florida
  - Tampa, Florida
  - Decatur, Georgia
  - Macon, Georgia
  - Chicago, Illinois
  - Baltimore, Maryland
  - Boston, Massachusetts
  - West Springfield, Massachusetts
  - Saint Louis, Michigan
  - Henderson, Nevada
  - Hillsborough, New Jersey
  - Santa Fe, New Mexico
  - Albany, New York
  - Manhasset, New York
  - New York, New York
  - Stony Brook, New York
  - The Bronx, New York
  - Durham, North Carolina
  - Huntersville, North Carolina
  - Hershey, Pennsylvania
  - Philadelphia, Pennsylvania
  - Memphis, Tennessee
  - Dallas, Texas
  - Houston, Texas
  - Annandale, Virginia
  - Seattle, Washington
  - Tacoma, Washington
- Santurce, Puerto Rico

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in the United States and Puerto Rico. The first participant was screened on 26 February 2007. The last study visit occurred on 24 March 2015.
Pre-assignment Details: Participants must have been enrolled in other Gilead-sponsored studies of elvitegravir (EVG) + ritonavir (RTV) to be eligible to receive continued access to EVG+RTV in this study.
Groups:
- EVG+RTV: Elvitegravir (EVG) 85 or 150 mg tablet boosted with ritonavir (RTV; r/) 100 mg capsule once daily with food in combination with an investigator-selected antiretroviral (ARV) regimen for the duration of the study.
  Some participants may have received EVG 300 mg during the course of protocol amendment 2.
Period: Overall Study
Arm/Group | EVG+RTV
Started | 192
Completed | 73
Not Completed | 119
Not completed — Withdrew Consent | 29
Not completed — Lack of Efficacy | 28
Not completed — Investigator's Discretion | 22
Not completed — Adverse Event | 13
Not completed — Lost to Follow-up | 13
Not completed — Death | 9
Not completed — Protocol Violation | 4
Not completed — Pregnancy | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: enrolled participants who received at least 1 dose of EVG
Groups:
- EVG+RTV: EVG 85 or 150 mg tablet boosted with RTV 100 mg capsule once daily with food in combination with an investigator-selected ARV regimen for the duration of the study. Some participants may have received EVG 300 mg during the course of protocol amendment 2.
Arm/Group | EVG+RTV
Number analyzed (Participants) | 192
Age, Continuous [Mean (Standard Deviation); unit: years] | 45 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 173
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 39
  Not Hispanic or Latino | 153
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Number; unit: participants]
  White | 139
  Black or African American | 48
  Native Hawaiian or Other Pacific Islander | 1
  Other | 4

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Experiencing Any Treatment-Emergent Study Dug-Related Adverse Event
Time Frame: Up to Week 408 plus 30 days
Population: Safety Analysis Set: enrolled participants who received at least 1 dose of EVG
Measure: Number; unit: percentage of participants
Arm/Group | EVG+RTV
Number analyzed (Participants) | 192
percentage of participants | 14.6

2. Secondary Outcome: Percentage of Participants Experiencing Treatment-Emergent Adverse Events
Description: Adverse events (AEs) occurring during treatment and for 30 days following the last dose of study drug were summarized across the participant population. A participant was counted once if they had a qualifying event.
Time Frame: Up to Week 408 plus 30 days
Population: Safety Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | EVG+RTV
Number analyzed (Participants) | 192
percentage of participants
  Any AE | 93.8
  Grade 3 or 4 AE | 45.3
  Grade 3 or 4 Drug-related AE | 3.1
  Serious AE | 44.8

3. Secondary Outcome: Percentage of Participants Experiencing Any Treatment-Emergent Laboratory Abnormality
Description: Treatment-emergent laboratory abnormalities were defined as values that increase at least one toxicity grade from baseline. The most severe graded abnormality from all tests was counted for each participant.
Time Frame: Up to Week 408 plus 30 days
Population: Participants in the Safety Analysis Set with at least 1 postbaseline measurement were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | EVG+RTV
Number analyzed (Participants) | 191
percentage of participants
  Grade 1 | 18.3
  Grade 2 | 31.9
  Grade 3 | 35.1
  Grade 4 | 14.1

4. Secondary Outcome: Percentage of Participants Experiencing Any Marked Treatment-Emergent Laboratory Abnormality
Description: A 'marked abnormality' was defined as a shift from grade 0 (or missing) at baseline to at least grade 3 postbaseline; or grade 1 at baseline to grade 4 postbaseline.
Time Frame: Up to Week 408 plus 30 days
Population: Participants in the Safety Analysis Set with at least 1 postbaseline measurement were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | EVG+RTV
Number analyzed (Participants) | 191
percentage of participants | 40.3

5. Secondary Outcome: Hemoglobin at Baseline and Change From Baseline at Weeks 24, 48, 96, 144, 192, 240, 288, 336, and 384
Time Frame: Baseline; Weeks 24, 48, 96, 144, 192, 240, 288, 336, and 384
Population: Participants in the Safety Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | EVG+RTV
Number analyzed (Participants) | 192
g/dL
  Baseline (n = 190) | 14.2 (1.86)
  Change at Week 24 (n = 165) | 0.1 (1.01)
  Change at Week 48 (n = 151) | 0.3 (1.12)
  Change at Week 96 (n = 139) | 0.2 (1.44)
  Change at Week 144 (n = 118) | 0.2 (1.40)
  Change at Week 192 (n = 106) | 0.3 (1.36)
  Change at Week 240 (n = 91) | 0.2 (1.54)
  Change at Week 288 (n = 84) | 0.3 (1.79)
  Change at Week 336 (n = 78) | 0.3 (1.49)
  Change at Week 384 (n = 70) | 0.4 (1.55)

6. Secondary Outcome: Red Blood Cell (RBC) Count at Baseline and Change From Baseline at Weeks 24, 48, 96, 144, 192, 240, 288, 336, and 384
Time Frame: Baseline; Weeks 24, 48, 96, 144, 192, 240, 288, 336, and 384
Population: Participants in the Safety Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: 10^6 cells/μL
Arm/Group | EVG+RTV
Number analyzed (Participants) | 192
10^6 cells/μL
  Baseline (n = 190) | 4.6 (0.65)
  Change at Week 24 (n = 165) | 0.0 (0.37)
  Change at Week 48 (n = 151) | 0.0 (0.35)
  Change at Week 96 (n = 139) | 0.0 (0.45)
  Change at Week 144 (n = 118) | 0.0 (0.50)
  Change at Week 192 (n = 106) | 0.0 (0.48)
  Change at Week 240 (n = 91) | 0.0 (0.55)
  Change at Week 288 (n = 84) | 0.0 (0.55)
  Change at Week 336 (n = 78) | 0.0 (0.44)
  Change at Week 384 (n = 70) | 0.0 (0.45)

7. Secondary Outcome: White Blood Cell (WBC) Count at Baseline and Change From Baseline at Weeks 24, 48, 96, 144, 192, 240, 288, 336, and 384
Time Frame: Baseline; Weeks 24, 48, 96, 144, 192, 240, 288, 336, and 384
Population: Participants in the Safety Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: 10^3 cells/μL
Arm/Group | EVG+RTV
Number analyzed (Participants) | 192
10^3 cells/μL
  Baseline (n = 190) | 5.64 (2.074)
  Change at Week 24 (n = 165) | 0.02 (1.670)
  Change at Week 48 (n = 151) | 0.12 (1.899)
  Change at Week 96 (n = 139) | -0.17 (1.761)
  Change at Week 144 (n = 118) | -0.25 (1.948)
  Change at Week 192 (n = 106) | -0.19 (2.072)
  Change at Week 240 (n = 91) | -0.09 (2.082)
  Change at Week 288 (n = 84) | -0.21 (2.091)
  Change at Week 336 (n = 78) | -0.35 (1.961)
  Change at Week 384 (n = 70) | -0.28 (1.759)

8. Secondary Outcome: Platelet Count at Baseline and Change From Baseline at Weeks 24, 48, 96, 144, 192, 240, 288, 336, and 384
Time Frame: Baseline; Weeks 24, 48, 96, 144, 192, 240, 288, 336, and 384
Population: Participants in the Safety Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: 10^3 cells/µL
Arm/Group | EVG+RTV
Number analyzed (Participants) | 192
10^3 cells/µL
  Baseline (n = 187) | 226 (75.0)
  Change at Week 24 (n = 154) | 2 (47.3)
  Change at Week 48 (n = 148) | 5 (49.5)
  Change at Week 96 (n = 134) | 13 (59.4)
  Change at Week 144 (n = 114) | 3 (48.7)
  Change at Week 192 (n = 103) | -2 (53.8)
  Change at Week 240 (n = 88) | 6 (45.7)
  Change at Week 288 (n = 80) | 6 (60.9)
  Change at Week 336 (n = 76) | -6 (61.0)
  Change at Week 384 (n = 70) | -15 (56.8)

9. Secondary Outcome: Alkaline Phosphatase at Baseline and Change From Baseline at Weeks 24, 48, 96, 144, 192, 240, 288, 336, and 384
Time Frame: Baseline; Weeks 24, 48, 96, 144, 192, 240, 288, 336, and 384
Population: Participants in the Safety Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | EVG+RTV
Number analyzed (Participants) | 192
U/L
  Baseline (n = 192) | 101 (43.3)
  Change at Week 24 (n = 170) | -6 (26.8)
  Change at Week 48 (n = 156) | -9 (31.0)
  Change at Week 96 (n = 143) | -9 (28.9)
  Change at Week 144 (n = 122) | -13 (27.8)
  Change at Week 192 (n = 110) | -18 (27.7)
  Change at Week 240 (n = 95) | -17 (29.2)
  Change at Week 288 (n = 86) | -20 (29.3)
  Change at Week 336 (n = 80) | -19 (31.3)
  Change at Week 384 (n = 72) | -20 (33.5)

10. Secondary Outcome: Alanine Aminotransferase (ALT) at Baseline and Change From Baseline at Weeks 24, 48, 96, 144, 192, 240, 288, 336, and 384
Time Frame: Baseline; Weeks 24, 48, 96, 144, 192, 240, 288, 336, and 384
Population: Participants in the Safety Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | EVG+RTV
Number analyzed (Participants) | 192
U/L
  Baseline (n = 191) | 28 (16.6)
  Change at Week 24 (n = 169) | 2 (16.3)
  Change at Week 48 (n = 154) | 1 (17.5)
  Change at Week 96 (n = 141) | 2 (19.4)
  Change at Week 144 (n = 120) | 2 (18.6)
  Change at Week 192 (n = 109) | 1 (16.2)
  Change at Week 240 (n = 94) | 0 (18.0)
  Change at Week 288 (n = 85) | 3 (17.0)
  Change at Week 336 (n = 79) | 3 (22.9)
  Change at Week 384 (n = 71) | 1 (15.9)

11. Secondary Outcome: Aspartate Aminotransferase (AST) at Baseline and Change From Baseline at Weeks 24, 48, 96, 144, 192, 240, 288, 336, and 384
Time Frame: Baseline; Weeks 24, 48, 96, 144, 192, 240, 288, 336, and 384
Population: Participants in the Safety Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | EVG+RTV
Number analyzed (Participants) | 192
U/L
  Baseline (n = 185) | 29 (14.5)
  Change at Week 24 (n = 163) | 2 (13.4)
  Change at Week 48 (n = 150) | 0 (13.5)
  Change at Week 96 (n = 137) | 2 (16.2)
  Change at Week 144 (n = 116) | 1 (14.5)
  Change at Week 192 (n = 105) | -1 (12.4)
  Change at Week 240 (n = 91) | 0 (16.3)
  Change at Week 288 (n = 82) | 1 (12.8)
  Change at Week 336 (n = 76) | 1 (13.2)
  Change at Week 384 (n = 68) | 1 (12.0)

12. Secondary Outcome: HIV-1 RNA at Baseline and Change From Baseline at Weeks 24, 48, 96, 144, 192, 240, 288, 336, and 384
Time Frame: Baseline; Weeks 24, 48, 96, 144, 192, 240, 288, 336, and 384
Population: Participants in the Efficacy Analysis Set (enrolled participants who received at least 1 dose of EVG and had at least 1 postbaseline HIV-1 RNA or CD4 cell count measurement) with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | EVG+RTV
Number analyzed (Participants) | 191
log10 copies/mL
  Baseline (n = 190) | 2.70 (1.337)
  Change at Week 24 (n = 174) | -0.13 (0.795)
  Change at Week 48 (n = 158) | -0.20 (0.892)
  Change at Week 96 (n = 142) | -0.11 (0.963)
  Change at Week 144 (n = 123) | -0.22 (0.998)
  Change at Week 192 (n = 110) | -0.21 (1.043)
  Change at Week 240 (n = 96) | -0.15 (0.955)
  Change at Week 288 (n = 86) | -0.34 (1.066)
  Change at Week 336 (n = 82) | -0.70 (1.055)
  Change at Week 384 (n = 73) | -0.68 (1.029)

13. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 400 Copies/mL at Baseline and at Weeks 24, 48, 96, 144, 192, 240, 288, 336, and 384
Time Frame: Baseline; Weeks 24, 48, 96, 144, 192, 240, 288, 336, and 384
Population: Participants in the Efficacy Analysis Set with available data were analyzed. The missing-equals-excluded approach where participants with missing data were excluded from the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | EVG+RTV
Number analyzed (Participants) | 191
percentage of participants
  Baseline (n = 190) | 65.3
  Week 24 (n = 175) | 69.7
  Week 48 (n = 159) | 78.6
  Week 96 (n = 142) | 76.8
  Week 144 (n = 123) | 82.9
  Week 192 (n = 110) | 84.5
  Week 240 (n = 96) | 89.6
  Week 288 (n = 86) | 95.3
  Week 336 (n = 82) | 95.1
  Week 384 (n = 73) | 93.2

14. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL at Baseline and at Weeks 24, 48, 96, 144, 192, 240, 288, 336, and 384
Time Frame: Baseline; Weeks 24, 48, 96, 144, 192, 240, 288, 336, and 384
Population: as for outcome 13
Measure: Number; unit: percentage of participants
Arm/Group | EVG+RTV
Number analyzed (Participants) | 191
percentage of participants
  Baseline (n = 190) | 44.2
  Week 24 (n = 175) | 56.0
  Week 48 (n = 159) | 62.9
  Week 96 (n = 142) | 65.5
  Week 144 (n = 123) | 73.2
  Week 192 (n = 110) | 79.1
  Week 240 (n = 96) | 78.1
  Week 288 (n = 86) | 89.5
  Week 336 (n = 82) | 86.6
  Week 384 (n = 73) | 90.4

15. Secondary Outcome: CD4 Cell Count at Baseline and Change From Baseline at Weeks 24, 48, 96, 144, 192, 240, 288, 336, and 384
Time Frame: Baseline; Weeks 24, 48, 96, 144, 192, 240, 288, 336, and 384
Population: Participants in the Efficacy Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: cells/mm^3
Arm/Group | EVG+RTV
Number analyzed (Participants) | 191
cells/mm^3
  Baseline (n = 189) | 283 (211.8)
  Change at Week 24 (n = 168) | 22 (98.9)
  Change at Week 48 (n = 152) | 38 (119.5)
  Change at Week 96 (n = 138) | 78 (132.3)
  Change at Week 144 (n = 118) | 126 (177.0)
  Change at Week 192 (n = 106) | 149 (167.5)
  Change at Week 240 (n = 93) | 176 (198.1)
  Change at Week 288 (n = 84) | 205 (210.8)
  Change at Week 336 (n = 80) | 225 (206.8)
  Change at Week 384 (n = 71) | 234 (214.4)

16. Secondary Outcome: Incidence of Mortality
Description: The percentage of participants who died was summarized.
Time Frame: Up to Week 408 plus 30 days
Population: Safety Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | EVG+RTV
Number analyzed (Participants) | 192
percentage of participants | 6.8

ADVERSE EVENTS:
Time Frame: Baseline through end of study drug treatment (average exposure: 237 weeks) plus 30 days
Description: Safety Analysis Set: enrolled participants who received at least 1 dose of EVG
Groups:
- EVG+RTV: EVG 85 or 150 mg tablet boosted with RTV 100 mg capsule administered orally once daily with food in combination with an investigator-selected antiretroviral (ARV) regimen for the duration of the study.
  Some participants may have received EVG 300 mg during the course of protocol amendment 2.
Arm/Group | EVG+RTV
Serious Adverse Events (participants affected / at risk) | 86/192
Other Adverse Events (participants affected / at risk) | 172/192
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | EVG+RTV (N=192)
Anaemia (Blood and lymphatic system disorders) | 2
Lymphadenitis (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 3
Aortic valve stenosis (Cardiac disorders) | 1
Arteriosclerosis coronary artery (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 5
Atrial flutter (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 2
Cardiac failure congestive (Cardiac disorders) | 2
Cardiomyopathy (Cardiac disorders) | 1
Congestive cardiomyopathy (Cardiac disorders) | 2
Coronary artery disease (Cardiac disorders) | 1
Ischaemic cardiomyopathy (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 4
Vertigo (Ear and labyrinth disorders) | 1
Necrotising retinitis (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Colitis (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Duodenal perforation (Gastrointestinal disorders) | 1
Faecal incontinence (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 1
Intestinal prolapse (Gastrointestinal disorders) | 1
Oesophagitis (Gastrointestinal disorders) | 1
Pancreatitis acute (Gastrointestinal disorders) | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Chest pain (General disorders) | 3
Perforated ulcer (General disorders) | 1
Pyrexia (General disorders) | 2
Cholecystitis (Hepatobiliary disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 1
Serum sickness-like reaction (Immune system disorders) | 1
Anal abscess (Infections and infestations) | 1
Appendicitis (Infections and infestations) | 2
Aspergillus infection (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 5
Cryptosporidiosis infection (Infections and infestations) | 1
Diabetic foot infection (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 4
HIV infection (Infections and infestations) | 1
HIV wasting syndrome (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 2
Herpes zoster disseminated (Infections and infestations) | 1
Influenza (Infections and infestations) | 3
Listeriosis (Infections and infestations) | 1
Localised infection (Infections and infestations) | 1
Meningitis aseptic (Infections and infestations) | 1
Meningitis cryptococcal (Infections and infestations) | 1
Mycobacterium avium complex infection (Infections and infestations) | 1
Oesophageal candidiasis (Infections and infestations) | 2
Pneumocystis jirovecii pneumonia (Infections and infestations) | 2
Pneumonia (Infections and infestations) | 9
Pneumonia streptococcal (Infections and infestations) | 1
Progressive multifocal leukoencephalopathy (Infections and infestations) | 1
Prostatic abscess (Infections and infestations) | 1
Pseudomembranous colitis (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 2
Pyelonephritis acute (Infections and infestations) | 1
Secondary syphilis (Infections and infestations) | 1
Sepsis (Infections and infestations) | 2
Sinusitis aspergillus (Infections and infestations) | 1
Subcutaneous abscess (Infections and infestations) | 1
Urethritis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Viral infection (Infections and infestations) | 1
Viral pericarditis (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1
Hip fracture (Injury, poisoning and procedural complications) | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 1
Weight decreased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 4
Fluid overload (Metabolism and nutrition disorders) | 1
Gout (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 4
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1
Castleman's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Ataxia (Nervous system disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Cervical radiculopathy (Nervous system disorders) | 1
Hepatic encephalopathy (Nervous system disorders) | 1
Parkinson's disease (Nervous system disorders) | 1
Presyncope (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 2
Syncope (Nervous system disorders) | 1
Transient ischaemic attack (Nervous system disorders) | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1
Confusional state (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 2
Homicidal ideation (Psychiatric disorders) | 1
Major depression (Psychiatric disorders) | 1
Mental disorder (Psychiatric disorders) | 1
Mental status changes (Psychiatric disorders) | 4
Suicidal ideation (Psychiatric disorders) | 1
Suicide attempt (Psychiatric disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 5
Chronic kidney disease (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Renal impairment (Renal and urinary disorders) | 1
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 1
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Paranasal cyst (Respiratory, thoracic and mediastinal disorders) | 1
Pharyngeal ulceration (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1
Skin reaction (Skin and subcutaneous tissue disorders) | 1
Aortic stenosis (Vascular disorders) | 1
Deep vein thrombosis (Vascular disorders) | 3
Hypertension (Vascular disorders) | 1
Hypertensive crisis (Vascular disorders) | 1
Hypotension (Vascular disorders) | 2
Venous stenosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | EVG+RTV (N=192)
Lymphadenopathy (Blood and lymphatic system disorders) | 17
Hypogonadism (Endocrine disorders) | 11
Abdominal pain (Gastrointestinal disorders) | 12
Constipation (Gastrointestinal disorders) | 13
Diarrhoea (Gastrointestinal disorders) | 49
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 22
Nausea (Gastrointestinal disorders) | 32
Vomiting (Gastrointestinal disorders) | 16
Fatigue (General disorders) | 29
Pyrexia (General disorders) | 17
Seasonal allergy (Immune system disorders) | 10
Bronchitis (Infections and infestations) | 40
Cellulitis (Infections and infestations) | 16
Folliculitis (Infections and infestations) | 12
Herpes simplex (Infections and infestations) | 10
Influenza (Infections and infestations) | 19
Nasopharyngitis (Infections and infestations) | 34
Onychomycosis (Infections and infestations) | 11
Otitis media (Infections and infestations) | 12
Pharyngitis (Infections and infestations) | 15
Sinusitis (Infections and infestations) | 50
Upper respiratory tract infection (Infections and infestations) | 62
Urinary tract infection (Infections and infestations) | 15
Viral infection (Infections and infestations) | 11
Weight decreased (Investigations) | 14
Decreased appetite (Metabolism and nutrition disorders) | 14
Hyperlipidaemia (Metabolism and nutrition disorders) | 10
Arthralgia (Musculoskeletal and connective tissue disorders) | 26
Back pain (Musculoskeletal and connective tissue disorders) | 33
Muscle spasms (Musculoskeletal and connective tissue disorders) | 13
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 15
Pain in extremity (Musculoskeletal and connective tissue disorders) | 24
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 16
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 19
Dizziness (Nervous system disorders) | 10
Headache (Nervous system disorders) | 24
Neuropathy peripheral (Nervous system disorders) | 13
Anxiety (Psychiatric disorders) | 22
Depression (Psychiatric disorders) | 34
Insomnia (Psychiatric disorders) | 25
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 10
Erectile dysfunction (Reproductive system and breast disorders) | 14
Cough (Respiratory, thoracic and mediastinal disorders) | 33
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 13
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 14
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 14
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 11
Rash (Skin and subcutaneous tissue disorders) | 15
Hypertension (Vascular disorders) | 16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years